CLINICAL TRIAL: NCT05799339
Title: Exploring Engagement and Opportunities to Optimize CAB-LA as Pre-exposure Prophylaxis (PrEP) for Women Who Inject Drugs
Brief Title: Optimizing CAB-LA as PrEP for Women Who Inject Drugs
Status: Completed | Type: Observational
Sponsor: Alexis Roth (Other)
Collaborators: ViiV Healthcare (Industry); University of Miami (Other); University of Michigan (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Alexis Roth, Associate Professor, Drexel University
Organization: Drexel University (Other)
Other Study IDs: 2105008584_ViiV
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Opioid Use; Trauma, Psychological
Keywords: PrEP; Preexposure Prophylaxis; WWID; Women who inject drugs; CAB-LA; Long-acting injectable cabotegravir
MeSH Terms: conditions — HIV Infections; Psychological Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to elicit information crucial for designing strategies to support engagement in cabotegravir, a long-acting injectable form of pre-exposure prophylaxis (PrEP) to reduce HIV risk among women who inject drugs (WWID), a population with high unmet need that has been understudied in all phases of PrEP research. The main questions this study aims to answer are:

1. How do WWID perceive long-acting injectable cabotegravir (CAB-LA) as a HIV prevention tool?
2. If and how their decisions to initiate CAB-LA as PrEP are informed by their experiences with other long-acting medications, experience with daily oral medications, and their personal circumstance (e.g., like housing or addition severity)?
3. Do PrEP outcomes (e.g., adherence) and engagement in care over time differ between WWID prescribed CAB-LA versus daily oral PrEP?

The sample for this study will be derived from and ongoing prospective trial of "TIARAS," a multi-component behavioral intervention designed to reduce HIV acquisition risk among women who inject drugs (see NCT05192434).

DETAILED DESCRIPTION:
This open-label community demonstration project draws from parent study TIARAS (NCT05192434), a multi-component behavioral intervention designed to reduce HIV acquisition risk among women who inject drugs (WWID). Participants are prescribed PrEP prior to enrollment based on consultation with their medical provider. They then simultaneously enroll in TIARAS and this observational study. Over six months, we will use data extracted from participant's electronic medical records to (1) describe CAB-LA and daily oral PrEP uptake among WWID and (2) assess for differences in adherence and persistence among WWID prescribed CAB-LA versus daily oral PrEP. All quantitative analyses will control for random group assignment in the TIARAS trial (NCT05192434). To understand uptake (primary outcome), we will purposively sample 20 WWID who were prescribed CAB and 20 prescribed daily oral PrEP. Participants will complete a semi-structured interview designed to explore their decision to initiate PrEP and the product-related attributes that influenced their decision, accounting for previous PrEP experience or use of long-acting injectable medications (e.g., birth control or MOUD), and examining how structural factors, like homelessness or medical mistrust influence decision-making. To understand persistence and adherence, at endline (six-months) we will purposively recruit 10 women who initiated CAB-LA who remained actively engaged in care and 10 who did not. We will also purposively recruit 10 women who initiated daily oral PrEP who remained actively engaged in care and 10 who did not. All participants will complete a semi-structured interview that explores facilitators and barriers to adherence and persistence (secondary outcomes). We will focus on strategies to increase engagement in care. Because previous research highlights the important influence of seasons of risk on PrEP outcomes (i.e., women are less interested in PrEP during periods of low perceived HIV risk such as during drug abstinence), we will examine how individual and structural factors influence PrEP persistence. Finally, should we find that >10% of the sample switches or discontinues a PrEP formulation over time, we will recruit a subset (n=15) to understand their decision-making process about switching.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative cisgender female
* age ≥ 18 years
* speaks/reads English
* reporting past 6 months day non-prescription injection drug use
* enrolled in the TIARAS trial (NCT05192434)

Exclusion Criteria:

• Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender females eligible
Study Population: Women who inject drugs
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | 6-months
  PrEP uptake will be operationalized as the number of participants who are prescribed (1) CAB-LA AND receive their first injection OR (2) daily oral tenofovir-based PrEP AND receive their first week of medication, as verified in the patient's electronic medical record (EMR).

SECONDARY OUTCOMES:
CAB-LA adherence | 6-months
  To assess PrEP adherence in women initiating long-acting injectable cabotegravir (CAB-LA), we will extract the dates of CAB-LA injections from participants' electronic medical records and will determine whether each follow-up CAB-LA injection occurred within recommended dosing windows according to Apretude prescribing information (+/- 7 days). In primary analysis, any injection occurring within the recommended dosing window will be considered adherent. Injections outside this dosing window will be considered non-adherent.
PrEP persistence | 6-months
  To describe PrEP persistence, we will calculate the proportion of days covered by a PrEP prescription over the 12-month study period, among those who initiate PrEP (see PrEP uptake). Dates and number of pills dispensed and/or date of each CAB-LA injection will be extracted from the EMR. Persistence will be operationalized as: (sum of days with an "active" PrEP prescription) ÷ (365 days) × 100.
Late injection | 6-months
  Any CAB-LA injection occurring outside of the dosing window (+/- 7 days of each scheduled injection) will be considered late. Dates of each injection will be extracted from the patient's electronic medical record.
CAB-LA restart (reinitation) | 6-months
  A restart (reinitation) will be defined as any CAB-LA injection occurring more than 4 weeks from when it was scheduled/due but within the 12-month study timeframe. Dates for each CAB-LAI injection will be extracted from the patient's electronic medical record.
PrEP product switching | 6-months
  We will describe patterns of switching between PrEP modalities over time among those who initiate CAB-LA (see PrEP uptake). For example, we will assess the number/proportion of women switching from daily oral PrEP to CAB-LA (or vice versa), the timing of when switching occurred (e.g., after one month of PrEP uptake), and the average number of switches per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis M Roth, PhD, MPH, Principal Investigator — Drexel University
Locations (1):
- Prevention Point Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to TIARAS ClinicalTrials.gov protocol and results description — https://clinicaltrials.gov/ct2/show/NCT05192434?term=Alexis+Roth&cond=HIV&draw=1&rank=2